CLINICAL TRIAL: NCT07057011
Title: Therapeutic Outcomes of Selective Serotonin Reuptake Inhibitors and Phosphodiesterase-5 Inhibitors Combination Therapy Versus Monotherapy in Premature Ejaculation Patients With the Serotonin Transporter Gene Polymorphism (SLC6A4)
Brief Title: Therapeutic Outcomes of Selective Serotonin Reuptake Inhibitors and Phosphodiesterase-5 Inhibitors Combination Therapy Versus Monotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed, Resident at Dermatology , venereology and andrology, Faculty of medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ٍSerotonin Reuptake Inhibitors
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Paroxetine; Tablets; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Drug Comination Therapy) (Active Comparator): Twenty patients with premature ejaculation , matching inclusion & exclusion criteria as mentioned before, will receive SSRI (paroxetine 20mg/day) + PDE5 inhibitor (sildenafil 25mg/day) for 3 months . Follow up clinically every 4 weeks for 12 weeks.
  Interventions: Drug: Paroxetine 20 Mg Oral Tablet
- Group B (Monotherapy) (Active Comparator): Twenty patients with premature ejaculation will receive SSRI (paroxetine 20mg/day) + placebo for 3 months . Follow up clinically every 4 weeks for 12 weeks.
  Interventions: Drug: Paroxetine 20 Mg Oral Tablet
- Group C (Control) (Active Comparator): Twenty healthy matched individuals will receive placebo + placebo for 3 months . Follow up clinically every 4 weeks for 12 weeks.
  Interventions: Drug: Paroxetine 20 Mg Oral Tablet

INTERVENTIONS:
Drug: Paroxetine 20 Mg Oral Tablet — to compare the safety and efficacy of paroxetine alone versus the combination of paroxetine and sildenafil in Premature Ejaculation Patients with genetic polymorphism in the serotonin transporter gene-linked polymorphic region.
  Other Names: sildenafil 25mg Oral Tablet; Placebo

SUMMARY:
Premature ejaculation (PE) is a prevalent male sexual dysfunction that affects as many as 20-30% of men regardless of age and ethnicity.The International Society for Sexual Medicine defines premature ejaculation as a male sexual dysfunction characterised by ejaculation that always or nearly always occurs before or within about 1 minute of vaginal penetration from the first sexual experience (lifelong premature ejaculation) or a clinically significant and bothersome reduction in latency time, often to about 3 minutes or less (acquired premature ejaculation), the inability to delay ejaculation on all or nearly all vaginal penetrations and with negative personal consequences include distress, bother, frustration, and avoidance of sexual intimacy.

DETAILED DESCRIPTION:
Oral intake of tricyclic antidepressants and selective serotonin reuptake inhibitors (SSRI) has emerged as effective for patients with PE whether or not these patients suffered from depression. Sildenafil, a phosphodiesterase-5 inhibitor (PDE5i), was tried for premature ejaculation, and in one study associated with paroxetine (a SSRI), with IELT (intravaginal ejaculation latency time) going from 0.35 to 4.5 min.

Serotonin (5-hydroxytryptamine, 5-HT) plays an important role at the level of the central nervous system in the complex regulatory mechanisms involved in ejaculation. In clinical practice, selective serotonin reuptake inhibitor (SSRI) antidepressants (e.g., paroxetine, fluoxetine and sertraline) and the tricyclic antidepressant clomipramine are widely used to treat lifelong PE, suggesting that 5-HT and SSRIs play roles in the pathophysiology and treatment of PE. In this group, paroxetine and sertraline are often used effectively to treat PE, although none of these agents have been officially recognized as treatments for this condition.

SSRIs increase synaptic 5-HT concentrations in the ejaculation-related areas of the central nervous system by blocking 5-HT transporters. The serotonin transporter (5-HTT) plays an important role in the clearance of synaptic 5-HT, thereby regulating presynaptic and postsynaptic 5-HT receptor stimulation. Human 5-HTT is encoded by a single gene (SLC6A4) on chromosome 17q12. A polymorphism in the transcribed region can be caused by a 44-bp insertion ('long allele' [L]) or deletion ('short allele' [S]).

The transcriptional activity of the L allele has been reported to be twice as high as the S allele. Theoretically, men with one or more S alleles for the 5-HTT have fewer functioning transporters and could therefore lead to a higher serotonergic neurotransmission. Consequently, it is postulated that men with SS genotype have longer IELT durations than men with LL genotype.In the literature, a variety of findings have been reported concerning the relationship between 5-HTT polymorphism and the SSRI response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PE: Men aged 18-60 years with a diagnosis of PE according to the International Society for Sexual Medicine (ISSM) criteria.
* Healthy controls: Men aged 18-60 years without a history of PE or other sexual dysfunctions.

Exclusion Criteria:

* Other sexual dysfunctions: Erectile dysfunction, delayed ejaculation, or other sexual disorders.
* Cardiovascular disease: history of cardiovascular disease, hypertension, or stroke.
* Neurological or psychiatric disorders: Conditions that may affect sexual function, such as depression, anxiety, or Parkinson's disease.
* Medications affecting sexual function: Current use of medications that may impact sexual function, such as antidepressants or antipsychotics.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Treatment of premature ejaculation | 3 months
  Treating the patients whom having Premature Ejaculation with selective serotonin reuptake inhibitors and Phosphodiesterase-5 Inhibitors Combination Therapy with genetic polymorphism in the serotonin transporter gene-linked polymorphic region.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Adam Ali El-Taib, Professor, Study Chair — Dermatology, venereology and andrology ,Qena Faculty of medicine ,south valley university.; Ebtehal Alaa El-Din Kotop Mohamed, Lecturer, Study Director — Dermatology, venereology and andrology ,Qena Faculty of medicine ,south valley university.
Locations (1):
- South Valley University Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No